CLINICAL TRIAL: NCT03175237
Title: Mirror Therapy: Technique Benefits in Different Motor Impairment in Post-stroke Subjects
Brief Title: Mirror Therapy in Pos Stroke Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Roberta de Oliveira Cacho, Roberta de Oliveira Cacho, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 262.686
Record Dates: First submitted 2017-05-20; First posted 2017-06-05 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of Motor Patterns (Experimental): For the mirror therapy protocol applied to the Motor Standard, each patient was treated with 15 mirror therapy sessions, 3 times a week for a total duration of 50 minutes. There were 4 exercises of voluntary range of motion involving the extension and mass flexion of the fingers, adduction and abduction of the fingers, pronation and supination of the forearm and elbow extension with associated shoulder elevation.
  Interventions: Other: Mirror Therapy
- Group of Functional Activities (Experimental): For the mirror therapy protocol applied to functional activities, four functional exercises were performed: fitting of pieces stimulating fine and thick gripping, stacking of cubes / cups and transfer of objects of different shapes and sizes. Each patient was treated with 15 mirror therapy sessions, 3 times a week with a total duration of 50 minutes
  Interventions: Other: Mirror Therapy

INTERVENTIONS:
Other: Mirror Therapy

SUMMARY:
To evaluate the benefits of Mirror Therapy (MT) and motivation in patients with different levels of post-stroke motor impairment with two different therapy protocols. This is a randomized uncontrolled blinded study, with 27 individuals in the chronic phase of stroke. Participants were randomized into two intervention groups: MT group with motor patterns of movement (MP, n=13) and MT group with specific functional activities (SA, n=14). Motor impairment assessments (Fugl-Meyer Assessment - FMA), motivation (Intrinsic Motivation Inventory) and functionality (Functional Independence Measure - FIM) were performed before and after treatment, and 3 months after the end of sessions (follow-up). In each intervention group,there were patients classified with mild, moderate or severe motor impairment, according to FMA. All participants performed 15 MT sessions, 3 times a week for 50 minutes each session.

DETAILED DESCRIPTION:
Objective: To evaluate the benefits of Mirror Therapy (MT) and motivation in patients with different levels of post-stroke motor impairment with two different therapy protocols. Methods: This is a randomized uncontrolled blinded study, with 27 individuals in the chronic phase of stroke. Participants were randomized into two intervention groups: MT group with motor patterns of movement (MP, n=13) and MT group with specific functional activities (SA, n=14). Motor impairment assessments (Fugl-Meyer Assessment - FMA), motivation (IntrinsicMotivationInventory) and functionality (Functional Independence Measure - FIM) were performed before and after treatment, and 3 months after the end of sessions (follow-up). In each intervention group,there were patients classified with mild, moderate or severe motor impairment, according to FMA. All participants performed 15 MT sessions, 3 times a week for 50 minutes each session.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were age over 18 years, clinical diagnosis of chronic and unilateral stroke (greater than six months after injury), hemiparesis sequel in the upper limb, absence of severe cognitive impairment with scores for the Mini Mental State Examination (MMSE) greater than or equal to 24 points for the educated and 14 for uneducated 17 and good sitting balance, qualified with scores between 20 and 40 on the Berg Balance Scale (BBS)

Exclusion Criteria:

* Those with other neurological diseases and associated physical or mental disabilities, stroke trauma, pain and joint contractures in the upper limb that prevented movement and the ones who missed therapy more than 3 times in a row were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-05-10 (Actual); Primary Completion 2015-08-15 (Actual); Study Completion 2015-09-30 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment Scale | baseline, 8 weeks and 3 months (follow-up)
  Sensory and motor Impairment in post-stroke subjects. Severity of motor damage. In this case, use only upper limb session (score 66)

SECONDARY OUTCOMES:
Mini-mental state examination | baseline
  brief assessment of cognition
Berg Balance Scale | baseline
  Assessment of the static, dynamic and anticipatory balance
Intrinsic Motivation Inventory | baseline, 7 days and 14 days
  self-report measure of intrinsic motivation
Functional Independence of measure | baseline, 8 weeks and 3 months (follow-up)
  Assessment of activities of daily living and social cognition

CONTACTS AND LOCATIONS:
Overall Officials: Roberta O Cacho, PhD, Principal Investigator — Universidade Federal do Rio Grande do Norte

IPD SHARING:
Plan to Share IPD: No